CLINICAL TRIAL: NCT06946719
Title: Comparison of Octenidine and Sodium Hypochlorite for Pulp Irrigation in Direct Pulp Capping
Brief Title: Octenidine and Sodium Hypochlorite for Pulp Irrigation in Direct Pulp Capping
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, cemre koç, Dr., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023/04
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pulp Exposure, Dental
Keywords: pulp exposure; calcium silicate cement
MeSH Terms: conditions — Dental Pulp Exposure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Octenidine (Experimental): A cotton pellet soaked in 0.1% Octenidine will be applied to the exposed pulp area
  Interventions: Other: pulp lavage Octenidine
- NaOCl (Experimental): A cotton pellet soaked in 2.5% NaOCl will be applied to the exposed pulp area
  Interventions: Other: pulp lavage NaOCl

INTERVENTIONS:
Other: pulp lavage Octenidine — Use of Octenidine as a pulp irrigation solution in pulp capping for mature permanent teeth
  Arms: Octenidine
Other: pulp lavage NaOCl — Use of NaOCl as a pulp irrigation solution in pulp capping for mature permanent teeth
  Arms: NaOCl

SUMMARY:
In the included patients, after complete removal of caries from the entire cavity, the exposed pulp will be treated with either a 2.5% NaOCl or 0.1% Octenidine solution. Subsequently, the cavity will be restored using calcium silicate cement, glass ionomer cement, and composite resin. Postoperatively, the patient's pain level will be assessed using the Visual Analogue Scale (VAS) at 24 and 72 hours, as well as on the 7th day. Responses to pulp sensitivity tests and periapical radiographs will be evaluated at 6 months.

DETAILED DESCRIPTION:
After obtaining a detailed pain history from the patients and conducting clinical and radiographic examinations, if a case is deemed suitable for the study, patients will be informed about the possibility of participating in this research project and the procedures involved. The risks and benefits associated with the study will be explained to the patients. Once a patient is considered a potential candidate for the study and expresses interest in participation, informed consent will be obtained.

Before the caries removal procedure, local anesthesia will be administered, and the teeth will be isolated using a rubber dam. Cavities will be prepared using a diamond bur under continuous water cooling. Caries will be completely removed from the entire cavity with the help of steel round burs and excavators, continuing until hard dentin is reached. Bleeding from the exposed pulp will be controlled by pressing a cotton pellet soaked in sterile physiological saline onto the exposure site for one minute. At this point, a researcher not involved in this study will provide the treating clinician with a glass dish containing either a 2.5% NaOCl or 0.1% Octenidine solution. A cotton pellet soaked in the test or control solution will be applied to the exposed pulp, and the cavity will be gently wiped. The cavity will be restored using calcium silicate cement, glass ionomer cement, and composite resin. Postoperatively, the patient's pain levels will be assessed using the Visual Analogue Scale (VAS) at 24 and 72 hours, as well as on the 7th day. Pulp sensitivity tests and periapical radiographs will be conducted at 6 months to evaluate the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic posterior tooth (premolar or molar) with deep caries
* A healthy periodontal status, normal probing depth, and restorable.
* Negative responses to percussion and palpation tests while responding positively to cold testing and electric pulp testing

Exclusion Criteria:

* Participants will be excluded if they had any systemic diseases
* A negative response to cold testing and electric pulp testing.
* Presence of a sinus tract, absence of pulp exposure following complete caries removal, or necrotic or partially necrotic pulp tissue

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 24 hours
  Use of the Visual Analog Scale (VAS) following the procedure
Post operative pain | 48 hours
  Use of the Visual Analog Scale (VAS) following the procedure
Post operative pain | 72 hours
  Use of the Visual Analog Scale (VAS) following the procedure

SECONDARY OUTCOMES:
Pulp vitality-ct | 6 months
  Evaluation through cold testing
Pulp vitality-ept | 6 months
  Evaluation through electric pulp testing
Pulp vitality-pr | 6 months
  Evaluation through periapical radiographic examinations

CONTACTS AND LOCATIONS:
Overall Officials: Cemre Koç, Principal Investigator — Aydın Adnan Menderes University, Faculty of Dentistry
Locations (1):
- Cemre Koç, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No